CLINICAL TRIAL: NCT00372801
Title: A Double-Blind, Randomised, Placebo-Controlled, Cross-Over Pilot Study to Investigate the Efficacy of Ibuprofen in Patients With Osteoarthritis of the Knee Following Administration of a Single Dose
Brief Title: Effectiveness Of Single Doses Of Ibuprofen In Patients With Osteoarthritis Of The Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: COX103843
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Ibuprofen; COX2; VAS; knee; single dose
MeSH Terms: conditions — Osteoarthritis | interventions — Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen

SUMMARY:
To demonstrate that new drugs work, many complex multidose studies are often required. The intent of this study is to use Ibuprofen as an example of a marketed pain relief drug to validate a simpler single dose model for future assessment of new pain drugs.

ELIGIBILITY:
Inclusion criteria:

* Subjects diagnosed with primary Osteoarthritis of the knee.
* Have at least 3 months in symptom duration prior to screening visit.
* Regular user of a prescribed non-steroidal anti-inflammatory drug (NSAID) or selective cyclo-oxygenase II (COX2) inhibitor for management of knee pain.
* Pain walking on flat surface within specific interval prior to study start.

Exclusion criteria:

* History of hypersensitivity to NSAIDS.
* Allergy to Ibuprofen.
* Use of assistive devices other than a cane or knee brace.
* History of specified diseases/illnesses.
* Abnormal blood tests pre-study.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Start 2005-08

PRIMARY OUTCOMES:
Pain intensity recorded over 0-8 hours using question 1 of the WOMAC (Western Ontario and McMaster University Osteoarthritis Index)pain subscale (visual analog scale).

SECONDARY OUTCOMES:
Responder rate Patient impression of change - 8 & 24 hrs post dose Time to use of rescue medication (paracetamol)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, Sydney, New South Wales, Australia